CLINICAL TRIAL: NCT02236273
Title: Comparative Effectiveness of Interactive, Health Literacy Promoting Text Messages on HPV Vaccine Completion In Minority Adolescents
Brief Title: Interactive, Health Literacy Promoting Text Messages and HPV Vaccine Completion In Minority Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Stockwell, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: AAAM3960
Record Dates: First submitted 2014-09-07; First posted 2014-09-10 (Estimated); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Human Papillomavirus
Keywords: Human papillomavirus; vaccination; text message; reminder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Conventional Text Message (Experimental): Conventional text message reminder
  Interventions: Behavioral: Conventional text message reminder
- Enhanced reminders (Experimental): Enhanced text message reminders
  Interventions: Behavioral: Enhanced text message reminders

INTERVENTIONS:
Behavioral: Conventional text message reminder — Receipt of conventional text message notifying when due for next dose
  Arms: Conventional Text Message
Behavioral: Enhanced text message reminders — Receipt of enhanced text messages notifying when due for next dose coupled with educational information
  Arms: Enhanced reminders

SUMMARY:
Emerging communication technologies, such as text messaging offer low-cost, scalable opportunities to improve health literacy and promote healthy behaviors, such as vaccination. While the investigators reported the success of text message vaccine reminders, effects were limited by their untailored approach. The trans-theoretical model of behavior change supports tailoring interventions to an individual's stage of decision-making. Human papillomavirus (HPV) is the most prevalent sexually transmitted virus in the U.S. and can lead to genital warts, and cervical, anal and penile cancer. The three-dose vaccine is 90-100% efficacious. Minorities are at greatest risk for such cancers but have low HPV vaccine completion rates. Limited health literacy regarding the vaccine can affect series completion. The investigators will compare the effects of enhancing text message vaccination reminders with interactive, vaccine health literacy-promoting information tailored to vaccine decision making-stage on HPV vaccine series completion. The effects of these messages represent a new paradigm in interactive health communications.

ELIGIBILITY:
Inclusion Criteria:

* Parenting adult of adolescent age 11-17 years
* Adolescent received 1st dose of HPV at a study site within the last 2 weeks.
* Eligible parent's cell phone has text message capability

Exclusion Criteria:

* Language other than English or Spanish only
* Parent already in the study
* Intends to move away from the New York City area in <12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 956 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wynn CS, Catallozzi M, Kolff CA, Holleran S, Meyer D, Ramakrishnan R, Stockwell MS. Personalized Reminders for Immunization Using Short Messaging Systems to Improve Human Papillomavirus Vaccination Series Completion: Parallel-Group Randomized Trial. JMIR Mhealth Uhealth. 2021 Dec 27;9(12):e26356. doi: 10.2196/26356. PMID 34958306

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Text Message | Enhanced Reminders
Started | 481 | 475
Completed | 481 | 475
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Text Message | Enhanced Reminders | Total
Number analyzed (Participants) | 481 | 475 | 956
Age, Customized [Count of Participants; unit: Participants]
  < 14 years | 443 | 437 | 880
  15- 17 years | 38 | 38 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 242 | 478
  Male | 245 | 233 | 478
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latinx | 270 | 255 | 525
  Black | 47 | 66 | 113
  White | 73 | 81 | 154
  Other | 91 | 73 | 164
Language [Count of Participants; unit: Participants]
  Spanish | 310 | 304 | 614
  English | 171 | 171 | 342

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed HPV Vaccine Series
Description: receipt of 3 doses of HPV vaccine by 12 months after initiation
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Text Message | Enhanced Reminders
Number analyzed (Participants) | 481 | 475
Participants | 364 | 344

2. Secondary Outcome: Time Between 1st and 2nd Dose
Description: Time elapsed in days between first and second dose- for those in need of three doses
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Conventional Text Message | Enhanced Reminders
Number analyzed (Participants) | 215 | 200
days | 84.1 (59) | 82.8 (57)

3. Secondary Outcome: Time Between 1st and 3rd Dose
Description: Time elapsed (in days) between 1st and 3rd dose for those in need of three doses
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Conventional Text Message | Enhanced Reminders
Number analyzed (Participants) | 178 | 156
days | 210 (43) | 210 (43)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Conventional Text Message | Enhanced Reminders
All-Cause Mortality (participants affected / at risk) | 0/481 | 0/475
Serious Adverse Events (participants affected / at risk) | 0/481 | 0/475
Other Adverse Events (participants affected / at risk) | 0/481 | 0/475

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT02236273/Prot_SAP_000.pdf